CLINICAL TRIAL: NCT01468883
Title: The Treatment of Stage I and II Carcinoma of the Breast With Mastectomy and Axillary Dissection vs. Excisional Biopsy Axillary Dissection, and Definitive Irradiation
Brief Title: The Treatment of Stage I and II Carcinoma of the Breast With Mastectomy and Axillary Dissection Versus Excisional Biopsy, Axillary Dissection, and Definitive Irradiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 790111; 79-C-0111; NCT00026845 (obsolete NCT alias)
Record Dates: First submitted 2011-10-01; First posted 2011-11-10 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Surgery; Radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M (Active Comparator): Modified radical mastectomy
  Interventions: Procedure: M
- X (Experimental): Excisional biopsy plus radiation
  Interventions: Radiation: X

INTERVENTIONS:
Procedure: M — Modified radical mastectomy
  Arms: M
Radiation: X — Excisional biopsy plus radiation
  Arms: X

SUMMARY:
Patients with biopsy proven breast cancer, clinical stage I and II, will be randomized to receive treatment by one of two methods: (1) total mastectomy and axillary dissection; or (2) excisional biopsy, axillary dissection, and definitive irradiation.

Data from single institutions and from retrospective comparisons suggest that definitive irradiation with cosmetically acceptable breast preservation offers survival and local control results equivalent to extirpative surgery. This study will test this hypothesis in a prospective, randomized manner. After primary therapy, subjects will be followed for: (1) survival; (2) sites of recurrence; (3) anatomic function; (4) complications of therapy; and (5) cosmesis.

DETAILED DESCRIPTION:
Patients with biopsy proven breast cancer, clinical stage I and II, will be randomized to receive treatment by one of two methods: (1) total mastectomy and axillary dissection; or (2) excisional biopsy, axillary dissection, and definitive irradiation.

Data from single institutions and from retrospective comparisons suggest that definitive irradiation with cosmetically acceptable breast preservation offers survival and local control results equivalent to extirpative surgery. This study will test this hypothesis in a prospective, randomized manner. After primary therapy, subjects will be followed for: (1) survival; (2) sites of recurrence; (3) anatomic function; (4) complications of therapy; and (5) cosmesis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Female patients of any age with a dominant breast mass meeting the following requirements are eligible for this protocol:

On clinical evaluation the tumor must be confined to the breast and axillary lymph nodes (stage I and II).

Biopsy of the tumor must be classified as a primary breast neoplasm of epithelial origin.

Patients must be geographically accessible for follow-up and willing to return for the follow-up at the NCI.

Patient must be mentally competent to understand and give informed consent for the protocol.

EXCLUSION CRITERIA:

Patients will be excluded from this protocol for the following reasons:

Advanced local disease or distant metastases (stage III and IV);

Inflammatory cancer;

Chronic diseases such as heart, lung, liver, kidney, blood, or metabolic disorders which may render the patient a poor operative risk;

History of another cancer other than skin cancer (non-melanoma);

Concurrent pregnancy or lactation;

Non-palpable lesions manifested only by nipple discharge or skin rash (Paget's disease);

Previous therapy to the breast cancer other than excisional biopsy;

Multiple masses or multiple suspicious areas on mammogram unless all but one are proven histologically benign; and

Bilateral breast carcinoma, either invasive or in-situ.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 1979-09-04 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Results of excisional biopsy followed by radiation therapy versus modified radiacal mastectomy | survival rate completion of study
  To compare the results of excisional biopsy followed by radiation therapy versus modified radiacal mastectomy

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1979-C-0111.html